CLINICAL TRIAL: NCT07179341
Title: Survival Nomogram for Patients With Thymic Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weijie Ye (Other)
Responsible Party: Sponsor-Investigator, Weijie Ye, Resident Doctor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2024-411-01
Record Dates: First submitted 2025-09-04; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Thymic Carcinoma
MeSH Terms: conditions — Thymoma | interventions — Thymectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training cohort (Active Comparator): 156 patients diagnosed with TC accepting surgery
  Interventions: Procedure: Thymectomy for thymic carcinoma
- Validation cohort one (Placebo Comparator): 80 patients range from June 1, 1996, to January 1, 2015 accepting surgery
  Interventions: Procedure: Thymectomy for thymic carcinoma
- Validation cohort two (Placebo Comparator): 76 patients range from January 2, 2015, to July 1, 2023 accepting surgery
  Interventions: Procedure: Thymectomy for thymic carcinoma

INTERVENTIONS:
Procedure: Thymectomy for thymic carcinoma — Thymectomy for thymic cancer

SUMMARY:
Background Thymic carcinoma (TC) is a rare and aggressive mediastinal malignancy with poor prognosis. Our study aimed to develop a nomogram to predict overall survival (OS) of TC patients.

Method A total of 156 patients confirmed TC between 1996 and 2023 were selected from our database. They were divided into training cohort, validation cohort one and validation cohort two. A nomogram was constructed based on the risk factors affecting prognosis using a Cox proportional hazards regression model. The discrimination and calibration of the nomogram were evaluated by C-index, AUC and curve of calibration. The three cohorts were divided into low-risk and high-risk subgroups.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of TC in patients should be confirmed through endoscopic tumor biopsy or surgery to obtain tumor tissue for pathological confirmation under light microscope, and even further confirmed through immunohistochemical staining.
* Patients should accept surgery and obtain complete postoperative pathological reports in order to assess Masaoka-Koga staging.
* Patients who accepted surgery should be followed up at least six months or reached the endpoint event.

Exclusion Criteria:

* The patient had two types of primary tumors concurrently including TC.
* The tumor in the thymus was not primary but metastatic, having originated from a different primary site.
* The patient did not obtain a complete pathological report after surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of accepting surgery until the date of final documented or date of death from any cause, whichever came first, assessed up to 325 months
  Overall survival (OS) is the length of time a patient lives after a diagnosis or the start of treatment for a disease, such as cancer

CONTACTS AND LOCATIONS:
Locations (1):
- 651 Dongfeng Road East, Yuexiu District, Guangzhou, P.R. China, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No